CLINICAL TRIAL: NCT06214507
Title: An Observational Study of Genetic Cardiomyopathy, Danon Disease
Brief Title: Danon Disease Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-NI-A501-0223
Record Dates: First submitted 2023-11-17; First posted 2024-01-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Danon Disease
Keywords: Danon Disease; LAMP2; Lysosome-associated membrane protein 2; Cardiomyopathy; X-linked
MeSH Terms: conditions — Glycogen Storage Disease Type IIb; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort
  Interventions: Other: No intervention
- Retrospective Cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this international observational study is to learn about the natural history of Danon disease in male patients (≥8 years of age) and female patients (8 to 50 years of age).

DETAILED DESCRIPTION:
This is an international observational study with both retrospective and prospective data collection. The study is designed to describe the natural history of Danon disease, a rare X-linked genetic disorder, and one of the most severe and penetrant forms of inherited cardiomyopathy. This study will collect data about the clinical course of Danon disease, including signs and symptoms, key clinical events, and the impact of the disease on quality of life as managed with the current standard of care. A hybrid (retrospective and prospective data collection) approach is being used to generate robust and longitudinal data. A subset of patients will be used as an External Control Arm for comparison to RP-A501 Trial participants.

ELIGIBILITY:
Prospective Cohort:

1. Documentation of a pathogenic or likely pathogenic variant of the LAMP2 gene by a CLIA-certified genetic testing laboratory
2. Patient or parent/legal guardian are capable and willing to provide signed informed consent
3. Age ≥ 8 years at enrollment

   Female Prospective Cohort:
4. Evidence of left ventricular hypertrophy in the 12 months prior to or at enrollment.

   Retrospective (only) Cohort:
5. Documentation of a pathogenic or likely pathogenic variant of the LAMP2 gene by a CLIA-certified genetic testing laboratory
6. Patient or parent/legal guardian are capable and willing to provide signed informed consent, as required by local regulations
7. Age ≥ 8 years at enrollment
8. Prior cardiac transplantation or prior mechanical circulatory support
9. At least 30 days of retrospective medical records available prior to cardiac transplantation or mechanical circulatory support

   Female Retrospective (only) Cohort:
10. Prior evidence of left ventricular hypertrophy.

Key Exclusion Criteria:

All Cohorts:

1. Concurrent enrollment in any other clinical investigation involving use of an investigational agent for any condition at time of enrollment to this study that could confound interpretation of this study
2. Previous treatment with a gene therapy

   Prospective Cohort:
3. Prior mechanical circulatory support at time of enrollment to this study
4. Prior cardiac transplantation at time of enrollment to this study

   Female patients:
5. Age >51 years at enrollment

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients 8 years of age and over, Female patients 8 to 50 years of age (at the point of enrollment) with confirmed Danon disease recruited from a range of applicable care settings.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Mass Index (LVMI) by echocardiogram | Month 12, 24, 36
  Evaluation of change over duration of follow up

SECONDARY OUTCOMES:
Cardiac biomarkers (hsTnI) | Month 12, 24, 36 (when available)
  Evaluation of change over duration of follow up
Cardiac biomarkers (NT-proBNP, BNP) | Month 12, 24, 36 (when available)
  Evaluation of change over duration of follow up
NYHA class | Month 12, 24, 36
  Evaluation of change over duration of follow up
KCCQ-12 | Month 12, 24, 36
  Evaluation of change over duration of follow up
PedsQL | Month 12, 24, 36
  Evaluation of change over duration of follow up
Event free survival with events defined as death, heart transplant, mechanical circulatory support (MCS) or heart failure hospitalization | Month 12, 24, 36
  Evaluation over duration of follow up
Six Minute Walk Test | Month 12, 24, 36
  This test measures the distance that a subject can quickly walk on a flat, hard surface in a period of 6 minutes.
CBC | At enrollment
  CBC with differential
Serum Chemistry | At enrollment
  Electrolytes
ECG | Month 12, 24, 36
  Twelve-lead ECGs are relevant to describe changes in cardiac rhythm that may further contextualize the clinical events/endpointsevents/endpoints
Serum chemistry | At enrollment
  Creatinine
Serum chemistry | At enrollment
  LDH
Serum chemistry | At enrollment
  BUN
Serum chemistry | At enrollment
  eGFR
Serum chemistry | At enrollment
  LFT
Anti-AAV9 titer | Month 12, 24, 36
  Change in antibody assay findings over time

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center/New York Presbyterian, New York, New York
  - Texas Children's Hospital, Houston, Texas
- German Heart Center Munich, München, Germany
- Sheba Medical Center, Ramat Gan, Israel
- Azienda Ospedaliero Universitaria, Florence, Italy
- Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain
- University College London - Great Ormond Street Institute of Child Health, London, United Kingdom